CLINICAL TRIAL: NCT02397798
Title: Improved Ability to Cope With Everyday Life Through a Person-centered Training Program in Elderly Patients With Rheumatoid Arthritis - PEP-walk Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEp-walk study
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Person-centered high-intense training three times a week under supervision (supervision two times a week) during 5 months
  Interventions: Behavioral: Person-centered high-intense training under supervision
- Control (Active Comparator): Introduction to health-enhancing physical activity, personalized exercise program to perform at home three times a week during 5 months
  Interventions: Behavioral: Personalized exercise program to perform at home

INTERVENTIONS:
Behavioral: Person-centered high-intense training under supervision — A person-centered training program including a person-centered high-intense aerobic / strength training
  Arms: Intervention
Behavioral: Personalized exercise program to perform at home — Introduction to health-enhancing physical activity, personalized exercise program to perform at home three times a week
  Arms: Control

SUMMARY:
The purpose of this study is to examine whether person-centered high-intense aerobic / strength training during five months reduces inflammation and disease activity, improve immune cell function, and increases muscle strength, fitness and ability of the individual independence in elderly patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion

* Patients 65 years or older with RA diagnosed according to the ACR / EULAR 1987/2010 criteria,
* disease duration 2 years or more,
* disease activity as measured by DAS28 <5.1

Exclusion

* Comorbidities, such as unstable coronary artery disease, uncontrolled cardiac arrhythmia, or uncontrolled high blood pressure, which prevents moderate to intense exercise.
* Joint surgery completed within 6 months prior to study entry.
* Ongoing training at moderate to high level 2 or more times per week

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Ability to manage daily activities as measured by the rheumatoid arthritis-specific measure of the Health Assessment Questionnaire (HAQ). | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- VastraGotaland, Gothenburg, Sweden

REFERENCES:
- [Derived] Andersson SEM, Lange E, Kucharski D, Svedlund S, Onnheim K, Bergquist M, Josefsson E, Lord JM, Martensson IL, Mannerkorpi K, Gjertsson I. Moderate- to high intensity aerobic and resistance exercise reduces peripheral blood regulatory cell populations in older adults with rheumatoid arthritis. Immun Ageing. 2020 May 16;17:12. doi: 10.1186/s12979-020-00184-y. eCollection 2020. PMID 32467712
- [Derived] Lange E, Kucharski D, Svedlund S, Svensson K, Bertholds G, Gjertsson I, Mannerkorpi K. Effects of Aerobic and Resistance Exercise in Older Adults With Rheumatoid Arthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2019 Jan;71(1):61-70. doi: 10.1002/acr.23589. PMID 29696812